CLINICAL TRIAL: NCT01239355
Title: A Phase II Study of MK-2206 in Patients With Advanced Hepatocellular Carcinoma Who Have Failed or Are Intolerant of One Prior Line of Anti-angiogenic Therapy
Brief Title: MK2206 in Treating Patients With Advanced Liver Cancer That Did Not Respond to Previous Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early termination for discouraging results
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02549; NCI-2011-02549 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000688549; CHNMC-PHII-105; PHII-105 (Other: City of Hope Comprehensive Cancer Center); 8752 (Other: CTEP); P30CA033572 (NIH); N01CM00038 (NIH)
Record Dates: First submitted 2010-11-10; First posted 2010-11-11 (Estimated); Results first posted 2015-10-05 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2013-03

CONDITIONS: Adult Hepatocellular Carcinoma; Advanced Adult Hepatocellular Carcinoma; Localized Non-Resectable Adult Liver Carcinoma; Recurrent Adult Liver Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — MK 2206

ARMS (1):
- Treatment (Akt inhibitor MK2206) (Experimental): Patients receive oral Akt inhibitor MK2206 on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Akt Inhibitor MK2206; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Akt Inhibitor MK2206 — Given PO
  Other Names: MK2206
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well MK2206 works in treating patients with advanced liver cancer that did not respond to previous therapy. MK2206 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the median progression-free survival in patients with advanced hepatocellular carcinoma treated with MK-2206 after failure of one prior line of anti-angiogenic therapy.

SECONDARY OBJECTIVES:

I. Evaluate the objective response rate (CR + PR). II. Evaluate the median overall survival. III. Evaluate the tolerability and toxicity profile of MK-2206 in this patient population.

IV. Explore, in a preliminary fashion, potential molecular predictors of efficacy.

OUTLINE:

Patients receive oral Akt inhibitor MK2206 on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 4 weeks and then every 3-6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable or metastatic HCC for which standard curative measures do not exist

  * The diagnosis of hepatocellular carcinoma should be based on at least one of the following:

    * The presence of one or more liver lesions, measuring >= 2 cm, with characteristic arterial enhancement and venous washout in the setting of liver cirrhosis and/or hepatitis B or C infection
    * The presence of liver lesion(s) with AFP >= 400
    * Tissue confirmation in the absence of either or both of the above
    * Tissue availability is desired and will be sought, but tissue availability is not mandated for accrual to the study
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension, and that has not been the target of local or regional therapy including transarterial chemoembolization, intra-arterial chemotherapy, ethanol, or RFA ablation
* One prior line of systemic anti-angiogenic therapy is required; this type of therapy includes, but is not restricted to, sorafenib, bevacizumab, sunitinib, or brivanib given as single agents or in combination with other agents
* No clinically evident ascites (minimal, medically controlled ascites detectable on imaging studies only is allowed)
* No Child-Pugh C cirrhosis or Child-Pugh B cirrhosis with more than 7 points
* No fibrolamellar carcinoma or any mixed variants of HCC with dominant fibrolamellar histology
* Patients with known brain metastases should be excluded from this clinical trial
* ECOG 0-1
* Life expectancy of greater than 3 months
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count > 1,000 mcL
* Platelets >= 70,000/mcL
* Total bilirubin =< 1.5 institutional upper limit of normal
* AST (SGOT)/ALT (SGPT) < 5 x institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min
* Serum albumin >= 2.8 g/dL
* Not pregnant or nursing
* Fertile patients must use two forms of contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
* Must agree to collection of correlative blood samples during the study
* No patients unable to swallow pills or diagnosed with a gastrointestinal disorder that is likely to interfere with the absorption of MK-2206 or with the patient's ability to take regular oral medication
* Patients with hyperglycemia should be well controlled on oral agents before the patient enters the trial
* Patients with HgbA1C levels >= 8% or fasting blood glucose >= 150 mg/dL are not eligible for this study
* Baseline QTcF > 450 msec (male) or QTcF> 470 msec (female) will exclude patients from entry on study
* Patients with hepatitis B infection, defined by a positive hepatitis B surface antigen test, should be on suppressive anti-viral therapy

  * Only the following anti-viral therapies are allowed while a patient is on study: tenofovir disoproxil fumarate and entecavir
  * Patients with hypothyroidism must be on a stable dose of thyroid replacement and be clinically euthyroid
* No esophageal or gastric variceal bleeding within the last 6 months

  * Patients with prior history of variceal bleeding must have had an upper endoscopy (EGD) with appropriate treatment of varices within 6 months prior to study entry
* No uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
* None of the following:

  * Uncontrolled hypertension (systolic BP > 150 or diastolic BP > 100 on two occasions within two weeks of beginning therapy on this protocol)
  * Myocardial infarction within 6 months
  * NYHA class > II
  * Clinically significant bradycardia related to underlying cardiac disease
  * Clinically significant bundle branch block related to underlying cardiac disease
* No patients with second primary cancer (except adequately treated nonmelanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumors including lymphomas without bone marrow involvement curatively treated with no evidence of disease for ≥ 5 years)

  * The exception to this criterion is prostate cancer treated definitively with surgery and/or radiation with normal PSA and no clinical evidence of residual or recurrent prostate cancer
* HIV-positive patients on combination antiretroviral therapy are ineligible
* No history of allergic reactions attributed to compounds of similar chemical orbiologic composition to MK-2206 or other agents used in the study
* No medications that cause QTc interval prolongation
* Any number of prior regional therapies with transarterial chemoembolization, intra-arterial chemotherapy, or ablative therapy is allowed

  * No more than 1 prior line of systemic therapy for advanced and/or unresectable disease
* No patients who have had anti-angiogenic therapy, chemotherapy, radiotherapy or regional therapy (such as transarterial chemoembolization, intra-arterial chemotherapy) within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier

  * Localized radiation for palliation (i.e., bony metastasis, etc.) given for < 3 days is allowed before therapy and is not subject to the 4-week waiting requirement
  * Local ablative therapy such as radiofrequency ablation or cryotherapy must have been completed more than 2 weeks prior to study entry
* Patients may not be receiving any other investigational or non-investigational agents or therapies directed at treating their hepatocellular carcinoma
* Patients may not be receiving any other investigational agents for any condition
* Patients receiving any medications or substances that are inhibitors or inducers of CYP3A4 are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony El-Khoueiry, MD, Principal Investigator — University of Southern California, Norris
Locations (22):
- United States (22):
  - Tower Cancer Research Foundation, Beverly Hills, California
  - City of Hope Medical Center, Duarte, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Oncology Care Associates PLLC, Saint Joseph, Michigan
  - Saint John's Mercy Medical Center, St Louis, Missouri
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Akt Inhibitor MK2206): Patients receive 200mg oral Akt inhibitor MK2206 on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Akt Inhibitor MK2206: Given PO
  Laboratory Biomarker Analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Akt Inhibitor MK2206)
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 65 [50 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Estimated using the product-limit method of Kaplan and Meier. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions (the sum must also demonstrate an absolute increase of at least 5 mm), or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Until disease progression or death, up to 26 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 15
Months | 1.7 [1.6 to 3.0]

2. Secondary Outcome: Objective Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective Response (OR) = CR + PR
Time Frame: Evaluated for response every 2 cycles (8 weeks) with confirmatory evaluation at least 4 weeks following initial documentation of objective response, up to 26 months
Measure: Number; unit: participants
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 15
participants | 0

3. Secondary Outcome: Overall Survival
Description: Survival will be estimated by the product-limit (Kaplan-Meier) estimator.
Time Frame: Until death, up to 26 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 15
Months | 6.1 [3.0 to 8.4]

ADVERSE EVENTS:
Time Frame: Adverse events recorded over a period of 1 year and 5 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Treatment (Akt Inhibitor MK2206)
Serious Adverse Events (participants affected / at risk) | 6/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Akt Inhibitor MK2206) (N=15)
Ascites (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Movements involuntary (Nervous system disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Akt Inhibitor MK2206) (N=15)
Anemia (Blood and lymphatic system disorders) | 11 (17)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Bloating (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (6)
Diarrhea (Gastrointestinal disorders) | 6 (6)
Dry mouth (Gastrointestinal disorders) | 5 (6)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (3)
Mucositis oral (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (4)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Edema limbs (General disorders) | 2 (2)
Edema trunk (General disorders) | 1 (1)
Fatigue (General disorders) | 9 (14)
Fever (General disorders) | 2 (3)
Flu like symptoms (General disorders) | 2 (2)
Pain (General disorders) | 2 (2)
Mucosal infection (Infections and infestations) | 1 (1)
Activated partial thromboplastin time pr (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 7 (14)
Alkaline phosphatase increased (Investigations) | 8 (21)
Aspartate aminotransferase increased (Investigations) | 11 (26)
Blood bilirubin increased (Investigations) | 3 (11)
Creatinine increased (Investigations) | 3 (3)
Electrocardiogram QT corrected interval (Investigations) | 3 (6)
INR increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (7)
Neutrophil count decreased (Investigations) | 4 (6)
Platelet count decreased (Investigations) | 6 (17)
Weight gain (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 3 (11)
Anorexia (Metabolism and nutrition disorders) | 4 (5)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 9 (19)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (10)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (4)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (2)
Headache (Nervous system disorders) | 2 (4)
Presyncope (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (11)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (12)
Hypertension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated early after the first stage of a two-stage design, allowing for early termination for discouraging results

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less